CLINICAL TRIAL: NCT06789445
Title: A Phase 1/2a Study of Subretinal Administration of OpCT-001 Photoreceptor Precursor Cells Derived From iPSCs in Patients With Primary Photoreceptor Disease
Brief Title: A Study to Investigate the Safety of OpCT-001 in Adults Who Have Primary Photoreceptor Disease (CLARICO)
Acronym: CLARICO
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BlueRock Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: OpCT-001-101
Record Dates: First submitted 2025-01-17; First posted 2025-01-23 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Primary Photoreceptor Disease; Retinitis Pigmentosa (RP); Usher Syndrome; Cone-Rod Dystrophy; Inherited Retinal Disease (IRD); Rod-Cone Dystrophy; Rod-Cone Disease; Cone-Rod Disease; Retinal Degeneration
Keywords: Primary Photoreceptor disease; CLARICO; Photoreceptor cells; Inherited retinal disease; Cell Therapy; Cellular Therapy; Usher Syndrome; Cone-Rod Disease; Rod-Cone Disease; Retinitis Pigmentosa
MeSH Terms: conditions — Retinitis Pigmentosa; Usher Syndromes; Cone-Rod Dystrophies; Retinal Degeneration

STUDY DESIGN:
Intervention Model Description: Phase 1 of the study will include up to 4 planned dose levels to be administered across up to 4 cohorts. Phase 2 is planned to enroll a maximum of 15 participants per cohort in 2 cohorts to evaluate 2 dose levels of OpCT-001 that will be selected based on the Phase 1 safety and tolerability data.
Masking Description: Phase 1: None (Open Label) Phase 2: Investigator/study site personnel outside of the surgical team will be masked to dose level assignments
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Experimental): OpCT-001 dose level 1 will be administered via subretinal injection.
  Interventions: Biological: OpCT-001
- Cohort 2 (Experimental): OpCT-001 dose level 2 will be administered via subretinal injection.
  Interventions: Biological: OpCT-001
- Cohort 3 (Experimental): OpCT-001 dose level 3 will be administered via subretinal injection.
  Interventions: Biological: OpCT-001
- Cohort 4 (Experimental): OpCT-001 dose level 4 will be administered via subretinal injection.
  Interventions: Biological: OpCT-001

INTERVENTIONS:
Biological: OpCT-001 — Cell therapy product composed of photoreceptor precursor cells derived from human induced pluripotent stem cells (iPSCs).
  Arms: Cohort 1
Biological: OpCT-001 — Cell therapy product composed of photoreceptor precursor cells derived from human iPSCs.
  Arms: Cohort 2; Cohort 3; Cohort 4

SUMMARY:
Study OpCT-001-101 is a Phase 1/2a first-in-human, multisite, 2-part interventional study to evaluate the safety, tolerability, and the effect on clinical outcomes of OpCT-001 in up to approximately 54 adults with primary photoreceptor (PR) disease. Phase 1 will focus on safety and features a dose-escalation design. Phase 2 is designed to gather additional safety data and assess the effect of OpCT-001 on measures of visual function, functional vision, and anatomic measures of engraftment in different clinical subgroups.

DETAILED DESCRIPTION:
Phase 1 of the study will include up to 4 planned dose levels to be administered across up to 4 cohorts. Participants will be assigned to receive OpCT-001.

Dose escalation in Phase 1 will be conducted using a standard 3+3 scheme in which a total of up to 24 legally blind participants (~3 to 6 per cohort) will receive OpCT-001. Phase 2 is planned to enroll a maximum of 15 participants per cohort in 2 cohorts to evaluate 2 dose levels of OpCT-001 that will be selected based on Phase 1 safety and tolerability data. Phase 2 participants will be randomized 1:1 to either cohort. Phase 2 participants and the investigator/study site personnel outside of the surgical team will be masked to OpCT-001 dose assignments.

ELIGIBILITY:
Key Inclusion Criteria:

* Confirmed genetic diagnosis of primary photoreceptor (PR) disease
* Best corrected visual acuity (BCVA) in the study eye at Screening for Phase 1: Logmarithm of the minimum angle of resolution (LogMAR) 3.9 to LogMAR 1.0. BCVA at Screening for Phase 2: ETDRS letter score 20 and 60.
* Retinal structure examination in the study eye demonstrating regions suitable for cell administration.

Key Exclusion Criteria:

* History of/currently active clinically relevant, ocular inflammation or infection
* Glaucoma or other significant optic neuropathy
* Diabetic macular edema or diabetic retinopathy
* Clinically significant cystoid macular edema
* Spherical equivalent refractive error of greater than 8.00 diopters myopia
* Ocular surgery ≤3 months before Screening
* Monocular vision (ie, no light perception in the fellow eye)
* Presence of clinically significant anti-OpCT-001 Human Leukocyte Antigen (HLA) antibodies at Screening
* Currently active malignancy, or history of malignancy within 5 years before OpCT-001 administration. Exception: Basal cell carcinoma that has been definitively treated.
* Any current and active infection (bacterial/viral/fungal) that could put the participant at risk from immunosuppression
* History of any cell therapy, gene therapy, or retinal implant at any time
* Previously received a bone marrow or solid organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2029-10 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of ocular and non-ocular treatment-emergent adverse events (TEAEs) through the Week 52 visit | From OpCT administration through the Week 52 visit

SECONDARY OUTCOMES:
Change from baseline over time through the Week 52 visit in the treated portion of the study eye (SE) retina in outer retinal layer thickness as measured by spectral domain optical coherence tomography (SD-OCT) | From enrollment through the Week 52 visit

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Miami, Bascom Palmer Eye Institute, Miami, Florida
  - Retina Foundation of the Southwest, Dallas, Texas
  - University of Wisconsin, Madison, Wisconsin

REFERENCES:
- See also: Related Info — https://claricostudy.com/